CLINICAL TRIAL: NCT05893953
Title: Comparison of Spine Angle Between Immediate Feedback and Different Conditions of Normal Adult Seating Posture
Brief Title: Spine Angle Comparison in Adult Seating Posture With Immediate Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, JINHYUNG CHOI, Student, Sahmyook University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: sahmyook U
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Spinal Curvatures; Feedback, Psychological; Sitting Position
MeSH Terms: conditions — Spinal Curvatures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Healthy Students(Condition A) (Experimental): sitting in a standard chair wearing an immediately feedback device
  Interventions: Device: immediately feedback device
- Normal Healthy Students(Condition B) (Experimental): sitting in a gym-ball
  Interventions: Device: Unstable chair
- Normal Healthy Students(Condition C) (Experimental): sitting in a standard chair(control group)
  Interventions: Other: Standard chair

INTERVENTIONS:
Device: immediately feedback device — Sitting in a standard chair with immediate feedback device
  Arms: Normal Healthy Students(Condition A)
Device: Unstable chair — sitting in an unstable chair
  Other Names: gym-ball
  Arms: Normal Healthy Students(Condition B)
Other: Standard chair — Sitting in a standard chair
  Other Names: Control
  Arms: Normal Healthy Students(Condition C)

SUMMARY:
1. Background: In modern society, people are spending more time sitting due to the increased use of IT devices. Prolonged sitting with incorrect posture can lead to spinal deformities and an increase in spinal diseases. Common deformities include turtle neck posture, flat back, straight neck, and bent back. Misalignment of the spine is considered an important factor in causing spinal diseases, such as pain, arthritis, and degeneration. To address these issues, researchers have developed pillows and chairs that are ergonomically designed for everyday use and have been found to be effective.
2. Purpose: This study aims to investigate whether portable equipment can help individuals recognize and maintain correct sitting posture on their own.
3. Design: This study has a cross-sectional study design. Each condition is divided into three different sitting conditions. By using post-evaluation data, the intention is to compare the effects. (Condition A: sitting on a standard chair wearing an immediately feedback device, Condition B: sitting on a gym-ball, Condition C: sitting on standard chair)
4. Subject : Twenty-eight subjects were recruited as healthy students attending S University located in Nowon-gu, Seoul.
5. Result: The study found that maintaining a sitting posture immediately resulted in a statistically significant lower angle over time at the Cervicothoracic angle compared to other interventions. Similarly, a sitting posture immediately maintained a lower angle over time at the Thoracic angle compared to other sitting postures . However, the lumbar angle showed a significant increase over time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 20-year-olds with no visual and hearing problems and no problems with video viewing and agreeing to participate in the experiment

Exclusion Criteria:

* Those who needed treatment due to pain in the neck, chest, or back were excluded.

Those who had been diagnosed with a diagnosis that stopped studying and stopped sports activities in the past 12 months were excluded.

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Cervico-thoracic angle | 1minute, 5minute, 10minute
  Changes in the spine curvature in a sitting position over time
Thoracic angle | 1minute, 5minute, 10minute
  Changes in the spine curvature in a sitting position over time
Lumbar angle | 1minute, 5minute, 10minute
  Changes in the spine curvature in a sitting position over time

CONTACTS AND LOCATIONS:
Overall Officials: Choi Jinhyung, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook University, Seoul, Nowon-gu, South Korea